CLINICAL TRIAL: NCT05668065
Title: Immunogenicity of Heterologous Versus Homologous Prime Boost Schedule With mRNA and Inactivated COVID-19 Vaccines: a Single-blinded, Randomized, Parallel Group Superiority Trial
Brief Title: Immunogenicity of Heterologous Versus Homologous Prime Boost Schedule With mRNA and Inactivated COVID-19 Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Pasteur de Tunis (Other)
Responsible Party: Principal Investigator, Samar Samoud, Principal Investigator, Head of immunoallergology unit, Clinical Immunology Department, Institut Pasteur de Tunis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TN2021-NAT-INS-70
Record Dates: First submitted 2022-12-27; First posted 2022-12-29 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: Vaccine; Immunogenicity; Heterologous prime-boost; Coronavac; Pfizer-BioNtech
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: Randomized simple-blinded comparative phase III clinical trial
Who Masked: Participant
Masking Description: Simple-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoronaVac/CoronaVac (Experimental): Biological: Coronavac Two doses at 21-day +/- 3 days. Each innoculation dose is 0.5 ml containing 600 SU in-house unit (equals to 3μg) of SARS-CoV-2 antigen.
  Interventions: Biological: CoronaVac/CoronaVac
- CoronaVac/BNT162b2 (Active Comparator): Biological: CoronaVac/BNT162b2 First dose of Coronavac. Each innoculation dose is 0.5 ml containing 600 SU in-house unit (equals to 3μg) of SARS-CoV-2 antigen.
  Second dose of BNT162b2 at 21-day +/- 3 days. Each dose of the Pfizer-BioNTech COVID-19 Vaccine is 0.3 ml. Each prefilled syringe contains 30 mcg of a nucleoside-modified messenger RNA (modRNA) encoding the viral spike (S) glycoprotein of SARS-CoV-2.
  Interventions: Biological: CoronaVac/BNT162b2

INTERVENTIONS:
Biological: CoronaVac/CoronaVac — Two doses at 21-day +/- 3 days. Each innoculation dose is 0.5 ml containing 600 SU in-house unit (equals to 3μg) of SARS-CoV-2 antigen.
  Arms: CoronaVac/CoronaVac
Biological: CoronaVac/BNT162b2 — First dose of Coronavac. Each innoculation dose is 0.5 ml containing 600 SU in-house unit (equals to 3μg) of SARS-CoV-2 antigen.
  Second dose of BNT162b2 at 21-day +/- 3 days. Each dose of the Pfizer-BioNTech COVID-19 Vaccine is 0.3 ml. Each prefilled syringe contains 30 mcg of a nucleoside-modified messenger RNA (modRNA) encoding the viral spike (S) glycoprotein of SARS-CoV-2
  Arms: CoronaVac/BNT162b2

SUMMARY:
This study is a randomized, simple-blinded comparative phase III clinical trial comparing the immunogenicity of two doses Coronovac to that of a first dose of Coronovac (Sinovac, Beijing, China) followed by a booster shot with the mRNA-based BNT162b2 SARS-CoV-2 vaccine (Comirnaty, Pfizer-BioNTech).

The purpose of this study is to evaluate the superiority, safety and immunogenicity of the heterologous prime-boost CoronaVac/BNT162b2 vaccination to the homologous CoronaVac/CoronaVac regimen.

DETAILED DESCRIPTION:
This study is a randomized simple-blinded comparative phase III clinical trial in COVID-19 vaccine naïve volunteers adults aged between 18 and 60 years. The purpose of this study is to evaluate the superiority, safety and immunogenicity of the heterologous prime-boost CoronaVac/BNT162b2 vaccination to the homologous CoronaVac/CoronaVac regimen. The study is conducted in four different sites located in the North of Tunisia.

A total of 240 eligible participants were included. Among them, the primary end point data were available for 100 participants randomly allocated to heterologous boost group versus 99 participants randomly allocated to homologous boost dose group.

Participants are assigned to receive either two injections of the CoronaVac vaccine (1st and 2nd vaccine), or CoronaVac as 1st dose and Pfizer as 2nd dose in 3 to 4 weeks interval.

A blood sample (5ml of the whole blood) is collected for each participant at the vaccination center before the first dose injection. After verifying the absence of a SARS-CoV-2 infection during the interrogation (a follow-up survey), a 2nd blood sample (5ml of whole blood) is taken for each participant at the vaccination center before the second dose injection. After the two injections, a 3rd blood sample (5ml of whole blood) will be taken for each participant between day 21 and day 35 after the second dose. Data collection and all samples are treated at Institute Pasteur of Tunis.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance to participate in the study.
* Age: 18-60 years old.

Non-inclusion criteria:

* Presence of disability (mainly mental disability).
* Pregnancy.
* Patients under immunosuppressive treatment or immunocompromised individuals.
* Prior Covid-19 infection.

Exclusion Criteria:

* Occurrence of a serious adverse event (death, anaphylactic shock, ...).
* Subjects wishing to withdraw from the study.
* Occurrence of a SARS-CoV-2 symptomatic infection during the follow-up period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Superiority of the heterologous prime-boost immunization with mRNA vaccine after vaccination with an inactivated vaccine versus homologous immunization with inactivated vaccines | Between day 21 and day 35 after the second dose of vaccination
  The primary end point for immunogenicity was the serum neutralizing antibody level with a percentage of inhibition at 90% at 21-35 days after boost. A difference of 25% between groups was considered clinically relevant.

SECONDARY OUTCOMES:
Immunogenicity parameters (Neutralizing antibody and IgG antibody titers) between day 21 and day 35 | Between day 21 and day 35 after the second dose of vaccination
  The level of neutralizing antibodies and anti-spike IgG antibody responses
Immunogenicity parameters (Neutralizing antibody and IgG antibody titers) at day 0 (at baseline) | At day 0 (at baseline)
  The level of neutralizing antibodies and anti-spike IgG antibody responses
Immunogenicity parameters (Neutralizing antibody and IgG antibody titers) at day 21 +/- 3 days | At day 21 +/- 3 days after the first dose of vaccination
  The level of neutralizing antibodies and anti-spike IgG antibody responses
Safety indexes of adverse reactions at day 30 | At day 30 after the second dose of vaccination
  The incidence of adverse reactions at day 30 of the second dose of vaccination

CONTACTS AND LOCATIONS:
Locations (5):
- Tunisia (5):
  - Leoni factory (Governorate of Bizerte), Bizerte, Mateur
  - Géant supermarket (Governorate of Ariana), Aryanah, Mnihla
  - Vaccination center of Ariana, Aryanah
  - STEG head office (Governorate of Tunis), Tunis
  - Institut Pasteur de Tunis, Tunis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanriover MD, Doganay HL, Akova M, Guner HR, Azap A, Akhan S, Kose S, Erdinc FS, Akalin EH, Tabak OF, Pullukcu H, Batum O, Simsek Yavuz S, Turhan O, Yildirmak MT, Koksal I, Tasova Y, Korten V, Yilmaz G, Celen MK, Altin S, Celik I, Bayindir Y, Karaoglan I, Yilmaz A, Ozkul A, Gur H, Unal S; CoronaVac Study Group. Efficacy and safety of an inactivated whole-virion SARS-CoV-2 vaccine (CoronaVac): interim results of a double-blind, randomised, placebo-controlled, phase 3 trial in Turkey. Lancet. 2021 Jul 17;398(10296):213-222. doi: 10.1016/S0140-6736(21)01429-X. Epub 2021 Jul 8. PMID 34246358
- [Background] Khoury DS, Cromer D, Reynaldi A, Schlub TE, Wheatley AK, Juno JA, Subbarao K, Kent SJ, Triccas JA, Davenport MP. Neutralizing antibody levels are highly predictive of immune protection from symptomatic SARS-CoV-2 infection. Nat Med. 2021 Jul;27(7):1205-1211. doi: 10.1038/s41591-021-01377-8. Epub 2021 May 17. PMID 34002089
- [Background] Souza WM, Amorim MR, Sesti-Costa R, Coimbra LD, Brunetti NS, Toledo-Teixeira DA, de Souza GF, Muraro SP, Parise PL, Barbosa PP, Bispo-Dos-Santos K, Mofatto LS, Simeoni CL, Claro IM, Duarte ASS, Coletti TM, Zangirolami AB, Costa-Lima C, Gomes ABSP, Buscaratti LI, Sales FC, Costa VA, Franco LAM, Candido DS, Pybus OG, de Jesus JG, Silva CAM, Ramundo MS, Ferreira GM, Pinho MC, Souza LM, Rocha EC, Andrade PS, Crispim MAE, Maktura GC, Manuli ER, Santos MNN, Camilo CC, Angerami RN, Moretti ML, Spilki FR, Arns CW, Addas-Carvalho M, Benites BD, Vinolo MAR, Mori MAS, Gaburo N, Dye C, Marques-Souza H, Marques RE, Farias AS, Diamond MS, Faria NR, Sabino EC, Granja F, Proenca-Modena JL. Neutralisation of SARS-CoV-2 lineage P.1 by antibodies elicited through natural SARS-CoV-2 infection or vaccination with an inactivated SARS-CoV-2 vaccine: an immunological study. Lancet Microbe. 2021 Oct;2(10):e527-e535. doi: 10.1016/S2666-5247(21)00129-4. Epub 2021 Jul 8. PMID 34258603
- [Background] Vacharathit V, Aiewsakun P, Manopwisedjaroen S, Srisaowakarn C, Laopanupong T, Ludowyke N, Phuphuakrat A, Setthaudom C, Ekronarongchai S, Srichatrapimuk S, Wongsirisin P, Sangrajrang S, Imsuwansri T, Kirdlarp S, Nualkaew S, Sensorn I, Sawaengdee W, Wichukchinda N, Sungkanuparph S, Chantratita W, Kunakorn M, Rojanamatin J, Hongeng S, Thitithanyanont A. CoronaVac induces lower neutralising activity against variants of concern than natural infection. Lancet Infect Dis. 2021 Oct;21(10):1352-1354. doi: 10.1016/S1473-3099(21)00568-5. Epub 2021 Aug 26. No abstract available. PMID 34454652
- [Background] Lim WW, Mak L, Leung GM, Cowling BJ, Peiris M. Comparative immunogenicity of mRNA and inactivated vaccines against COVID-19. Lancet Microbe. 2021 Sep;2(9):e423. doi: 10.1016/S2666-5247(21)00177-4. Epub 2021 Jul 16. No abstract available. PMID 34308395
- [Background] Shaw RH, Stuart A, Greenland M, Liu X, Nguyen Van-Tam JS, Snape MD; Com-COV Study Group. Heterologous prime-boost COVID-19 vaccination: initial reactogenicity data. Lancet. 2021 May 29;397(10289):2043-2046. doi: 10.1016/S0140-6736(21)01115-6. Epub 2021 May 12. No abstract available. PMID 33991480
- [Background] Borobia AM, Carcas AJ, Perez-Olmeda M, Castano L, Bertran MJ, Garcia-Perez J, Campins M, Portoles A, Gonzalez-Perez M, Garcia Morales MT, Arana-Arri E, Aldea M, Diez-Fuertes F, Fuentes I, Ascaso A, Lora D, Imaz-Ayo N, Baron-Mira LE, Agusti A, Perez-Ingidua C, Gomez de la Camara A, Arribas JR, Ochando J, Alcami J, Belda-Iniesta C, Frias J; CombiVacS Study Group. Immunogenicity and reactogenicity of BNT162b2 booster in ChAdOx1-S-primed participants (CombiVacS): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet. 2021 Jul 10;398(10295):121-130. doi: 10.1016/S0140-6736(21)01420-3. Epub 2021 Jun 25. PMID 34181880